CLINICAL TRIAL: NCT05081986
Title: Motor Plasticity Enhancement of Spaced iTBS Trains: a Randomized, Placebo-controlled, Crossover Trial of D-cycloserine.
Brief Title: Repeated iTBS Cycloserine Motor Plasticity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Alexander McGirr, Assistant Professor, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: REB21-0863
Record Dates: First submitted 2021-09-27; First posted 2021-10-18 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity | interventions — Transcranial Magnetic Stimulation; Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- D-cycloserine (Experimental): Participants will ingest a capsule containing 100mg of the antibiotic d-cycloserine one hour prior to receiving theta-burst stimulation (TBS; a patterned stimulation). Their baseline motor evoked potentials (MEP) will be recorded for 20 minutes prior to receiving the first TBS to the motor cortex and change in MEP amplitude will be measured following stimulation up to 60minutes later. They will then receive a second TBS to the motor cortex and change in MEP amplitude will again be measured following stimulation up to 60minutes later.
  Interventions: Device: Transcranial Magnetic Stimulation; Drug: Cycloserine
- Placebo (Placebo Comparator): Participants will ingest a capsule identical to that containing the study medication, however this capsule will contain a placebo. They will ingest this capsule one hour prior to receiving theta-burst stimulation (TBS; a patterned stimulation). Their baseline motor evoked potentials (MEP) will be recorded for 20 minutes prior to receiving the first TBS to the motor cortex and change in MEP amplitude will be measured following stimulation up to 60minutes later. They will then receive a second TBS to the motor cortex and change in MEP amplitude will again be measured following stimulation up to 60minutes later.
  Interventions: Device: Transcranial Magnetic Stimulation; Drug: Placebo Oral Tablet

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Single-pulse transcranial magnetic stimulation and theta-burst stimulation
Drug: Cycloserine — Cycloserine 100mg
  Arms: D-cycloserine
Drug: Placebo Oral Tablet — Placebo capsule matched to cycloserine capsule
  Arms: Placebo

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) is a modality for probing and altering brain function in humans non-invasively. The technology relies on the principles of electromagnetic induction, whereby magnetic fields have an associated electrical field. By intersecting two magnetic fields safely generated outside the head, one can induce a focal electrical current where the magnetic fields intersect in the brain, and this can depolarize cell membranes and impact brain activity.

A well investigated phenomenon in neuroscience is the principle of long term potentiation (LTP), and its converse long term depression (LTD), referring to the ability of neurons to increase or decrease their connection strength in an activity dependent manner. They do this through modifications to their electrochemical junctions, the synapses. We have previously used the motor system as a model system to study the impact D-Cycloserine, an NMDA receptor partial agonist, on synaptic plasticity after TMS.

Conventional therapeutic TMS is delivered once daily, however it is increasingly being delivered multiple times per day in an effort to speed treatment effects. It is unclear how adjunctive agents would impact these repeated stimulation designs.

Research Question:

Does the N-methyl-D-aspartate receptor partial agonist D-Cycloserine stabilize motor plasticity across multiple daily sessions of TMS?

DETAILED DESCRIPTION:
Objectives:

1. To recruit 20 participants into a cross-over trial. These participants will complete two study phases (active and placebo), and will not know whether they are taking a low-dose d-cycloserine capsule (100mg) or a placebo capsule at each of these phases.
2. To measure motor evoked potentials (MEP) in the hand in relation to magnetic stimulation of the motor cortex responsible for this muscle. These will be measured at baseline, and after receiving rTMS over the motor cortex.
3. To deliver intermittent theta-burst rTMS stimulation (TBS) to the FDI region of the motor cortex.
4. To measure the magnitude (and associated change from baseline) of the MEPs after rTMS at a fixed stimulus intensity, and using a range of stimuli to generate a stimulus response curve.
5. To repeat iTBS one hour later and measure the impact on MEPs.
6. To measure changes in performance on computerized cognitive tasks following ingestion of the blinded capsule.

Methods:

D-Cycloserine will be purchased from Parsolex and repackaged into 100mg placebo-controlled capsules by Script Pharmacy in Calgary.

1. We will recruit 20 participants aged 18-65 through community advertisement, carefully screened for exclusion factors related to rTMS and DCS.
2. Participants will be randomly assigned by random number sequence with allocation concealment to one of two first arms of the crossover study: a) placebo-DCS 100mg and b) DCS 100mg-placebo.
3. Participants will complete the QIDS-SR (Quick Inventory of Depressive Symptoms-Self Report), the BAI (Beck Anxiety Inventory), and the STAI (State Trait Anxiety Inventory).
4. Participants will take their blinded capsule at least 1 hour prior to TBS. (we anticipate that it will take approximately 30 minutes to do steps 5-7)
5. Electromyographic (EMG) electrodes will be positioned over the first dorsal interosseous (FDI) bilaterally. These are non-invasive electrodes that use an adhesive to stick to the skin.
6. Using neuronavigation in conjunction with an atlas brain, the M1 hand strip will be localized using single pulse TMS (MagPro X100).
7. Motor evoked potentials are measurements of muscle activation, in this case in response to TMS stimulation of the brain. We will use single pulse TMS to record the magnitude of responses. As a baseline, we will collect twenty single-pulse (120% resting motor threshold (RMT), 0.25Hz) MEPs every 5 minutes for the 15 minutes preceding TBS rTMS. We will also characterize the stimulus response curve at baseline by delivering single pulse TMS at stimulus intensities ranging from 100-150% resting motor threshold presented in random order.
8. TBS rTMS will be applied to the FDI 'hotspot'. TBS consists of 2s trains every 10s. Trains are composed of 3 pulses at 50Hz, 200ms intervals, 80% RMT. Total time 190s and 600 pulses.
9. After TBS, twenty MEPs will be acquired (single pulse, 120% RMT, 0.25Hz) every 5 minutes for the first 15 minutes after iTBS. A stimulus response curve will be acquired at 30 minutes and 60 minutes post iTBS.
10. One hour following TBS, a second train of TBS rTMS will be applied to the FDI 'hotspot'. TBS consists of 2s trains every 10s. Trains are composed of 3 pulses at 50Hz, 200ms intervals, 80% RMT. Total time 190s and 600 pulses.
11. After TBS, twenty MEPs will be acquired (single pulse, 120% RMT, 0.25Hz) every 5 minutes for the first 15 minutes after iTBS. A stimulus response curve will be acquired at 30 minutes and 60 minutes post iTBS.
12. During one of the breaks in the stimulation procedure, a brief, computerized neurocognitive assessment will take place after ingestion of the blinded capsule.
13. Participants will be asked if they believe they received the study medication or placebo in this first phase of the crossover trial.

This is study involves a crossover design, therefore after a minimum of 7 days the experiment will be repeated with the second blinded capsule.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy (absence of chronic medical conditions) individuals
2. Aged 18-65. The lower limit is justified by the absence of safety studies involving DCS in pediatric studies, and the upper limit is justified by the increasing prevalence of chronic illness.

Exclusion Criteria:

1. Allergy to cycloserine
2. Are currently pregnant, breast feeding or plan to become pregnant
3. Have an alcohol or substance use disorder within the last 3 months
4. Current psychiatric concerns
5. are at a significant risk of harm to themselves or others
6. Have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of epilepsy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than or equal to 5 minutes
7. Have concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
8. Have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
9. Conditions that may impair the ability to metabolize cycloserine including, but not limited to current Renal or Liver Disease.
10. Inability to refrain from alcohol use for 24 hours prior to each session and following each session.
11. Use of isoniazid or ethionamide
12. Are currently (or in the last 4 weeks) using any benzodiazepine, cyclopyrrolone, gabapentin/pregabalin or anticonvulsant due to the potential to limit rTMS efficacy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Stimulus Response Curve (SRC): Change in stability through repeated intermittent Theta Burst Stimulation (iTBS) | SRC will be administered at baseline, 30 minutes after first iTBS, 60 minutes after first iTBS, 30 minutes after second iTBS, and 60 minutes after second iTBS
  SRC will be characterized by collecting Motor evoked potentials (MEPs) at stimulus intensities ranging from 100-150% resting motor threshold, presented in random order. How the SRC will change following multiple rounds of iTBS will be assessed.

SECONDARY OUTCOMES:
Motor Evoked Potential (MEP): Amplitude Time Course | Collected at baseline, 15 minutes following first iTBS, and 15 minutes following second iTBS
  Change in the (electrical) amplitude of muscle responses to stimulation of the motor cortex will be recorded from the first dorsal interosseous muscle of the hand.
Change in Cognitive Function - THINC-it- PDQ-5 | Administered once during each crossover arm, at 30-minutes following first iTBS.
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The cognitive questionnaire is called the Perceived Deficits Questionnaire - 5 item scale (PDQ-5). The questionnaire assesses self perceived cognition by asking questions about attention/concentration, retrospective memory, prospective memory, and planning/organization.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-it- Choice Reaction Time | Administered once during each crossover arm, at 30-minutes following first iTBS.
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The first objective cognitive test is called "spotter" and measures choice reaction time by calculating the total time that elapses between the presentation of a stimulus and the occurrence of a response in a task that requires a participant to make one of two different responses depending on which stimuli is presented.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-it- Working Memory | Administered once during each crossover arm, at 30-minutes following first iTBS.
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The second objective cognitive test is called "Symbol Check" and is an n-back test. N-back tests measure working memory by presenting the subject with a sequence of stimuli, and the task consists of selecting the stimuli that was presented n steps earlier in the sequence.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-it- Digit Symbol Substitution | Administered once during each crossover arm, at 30-minutes following first iTBS.
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The third objective cognitive test is called "CodeBreaker" and is a Digit Symbol Substitution Test (DSST). DSST involves a key consisting of the numbers 1-6, each paired with a unique symbol. Below the key are a series of the numbers 1-6 in random order and repeated several times. Subjects must select the corresponding symbol as fast as possible. The number of correct symbols within the allowed time is measured.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Cognitive Function - THINC-it- Trail Making Test part B | Administered once during each crossover arm, at 30-minutes following first iTBS.
  Cognitive function will be assessed using the THINC-it brief cognitive assessment tool. THINC-it includes a summation of four objective cognitive tests and a subjective cognitive questionnaire.
  The fourth objective cognitive test is called "Trails" and is a version of the Trail Making Test part B (TMT-B). The subject is presented with numbers and letters in circles placed in random array on the screen. The subject must draw a line from one circle to the next in ascending order; however, s/he must alternate the circles with numbers in them and circles with letters in them (ie, 1-A-2-B-3-C etc). The TMT is a timed test and the goal is to complete the tests accurately and as quickly as possible.
  Total results from the THINC-it assessment indicate cognitive performance compared to healthy age-, sex- and education-matched individuals. Change between the two arms will be assessed.
Change in Implicit Suicidal Thoughts | Administered once during each crossover arm, at 30-minutes following first iTBS.
  Death Implicit Association Test (D-IAT) is a behavioral test that measures the strength of automatic (implicit) associations between concepts in people's minds relying on latency measures in a simple sorting task. The strength of an association between concepts of "death" and "ones self" is measured by the standardized mean difference score of the 'hypothesis-inconsistent' pairings and 'hypothesis-consistent' pairings.
  Change between the two arms will be assessed.

OTHER OUTCOMES:
Safety outcomes | Through study completion, on average 1 week
  Adverse events will be tracked and recorded
Side Effects | Participants will complete the TSES before and after the 3-hour stimulation session.
  Side effects will be tracked through the Toronto Side Effects Scale (TSES). The TSES is a self reported questionnaire that assesses incidence, frequency, and severity of central nervous system, gastrointestinal, and sexual side effects. TSES will be administered before and after TMS sessions, and change in side effects will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McGirr, MD, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wrightson JG, Cole J, Sohn MN, McGirr A. The effects of D-Cycloserine on corticospinal excitability after repeated spaced intermittent theta-burst transcranial magnetic stimulation: A randomized controlled trial in healthy individuals. Neuropsychopharmacology. 2023 Jul;48(8):1217-1224. doi: 10.1038/s41386-023-01575-7. Epub 2023 Apr 11. PMID 37041205